CLINICAL TRIAL: NCT06378853
Title: Risk Factors of Postoperative Complications and Survival Rate in Pancreatic Ductal Adenocarcinoma Patients Based on Body Compositions Measured by 3D CT Scan and Hematological Indicators
Brief Title: Risk Factors of Postoperative Complications and Survival Rate in Pancreatic Ductal Adenocarcinoma Patients
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Professor, Jinling Hospital, China
Other Study IDs: 2023DZKY-049-01
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; risk factors; postoperative complications; overall survival
MeSH Terms: conditions — Pancreatic Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
By evaluating the nutritional status of patients with pancreatic ductal adenocarcinoma (PDAC) admitted to Jinling Hospital, collecting relevant clinical data. we aim to conduct correlation analysis with patient clinical information, such as survival time, hospitalization time, nutritional status, hematological indicators, etc., in order to reveal the prognostic factors for overall survival and postoperative complications of PDAC patients.

DETAILED DESCRIPTION:
Personalized and accurate survival risk prognostication remains a significant challenge in pancreatic ductal adenocarcinoma (PDAC), despite extensive research on prognostic and predictive markers. Patients with PDAC are prone to muscle loss, fat consumption, and malnutrition, which is associated with inferior outcomes. This study investigated the use of three-dimensional (3D) anthropometric parameters derived from computed tomography (CT) scans and hematological indicators in relation to overall survival (OS) outcomes and postoperative complications in PDAC patients.

A retrospective analysis was conducted on patients with PDAC, all of whom had undergone pretreatment abdomen-pelvis CT scans. Automatic 3D measurements of subcutaneous and visceral fat volume, skeletal muscle volume, and skeletal muscle density (SMD) were assessed at the L3 vertebral level by an artificial intelligence assisted diagnosis system (HY Medical). Various indicators including TyG-BMI, nutritional indicators [geriatric nutritional risk index (GNRI) and prealbumin], and inflammation indicators [(C-reactive protein (CRP) and neutrophil to lymphocyte ratio (NLR)] were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* All eligible patients diagnosed with PDAC

Exclusion Criteria:

* 1) Suffering from chronic or acute diseases related to malnutrition: chronic heart failure, cirrhosis, chronic kidney disease and infection, cognitive impairment, dysphagia or gastrointestinal obstruction, etc; 2) Using excessive doses of systemic glucocorticoids within 4 weeks prior to enrollment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tumors of patients are histopathologically confirmed as PDAC
Sampling Method: Non-Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
complications | 2019/1/1-2023/12/31
  the postoperative complications in PDAC patients
overall survival | 2019/1/1-2023/12/31
  overall survival of PDAC patients
risk factors | 2019/1/1-2023/12/31
  risk factors of PDAC patients

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No